CLINICAL TRIAL: NCT04732455
Title: Intravenous Lidocaine Infusion Versus Oral Duloxetine For The Prevention And Treatment Of Chemotherapy Induced Peripheral Neuropathy Among Breast Cancer Patients
Brief Title: Lidocaine Versus Duloxetine for the Prevention of Taxane-Induced Peripheral Neuropathy In Breast Cancer Patients
Acronym: TIPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gamal Mohamed Taha Abouelmagd (Other)
Responsible Party: Sponsor-Investigator, Gamal Mohamed Taha Abouelmagd, MSc Anaesthesia and Surgical Intensive Care, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1216-4-011
Record Dates: First submitted 2021-01-16; First posted 2021-02-01 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Peripheral Neuropathy; Chemotherapy-induced Peripheral Neuropathy; Breast Cancer
Keywords: Breast cancer; Chemotherapy; Lidocaine; Duloxetine; Taxane induced peripheral neuropathy (TIPN)
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms | interventions — Lidocaine; Sodium Chloride; Duloxetine Hydrochloride; Fumigant 93; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Control (C) (Placebo Comparator): 20 adult breast cancer patients on Taxane chemo protocol will receive 200 ml normal saline over forty minutes pre each chemotherapy session until end of the cycle.
  Interventions: Drug: Normal saline
- Group lidocaine infusion (L) (Experimental): 20 adult breast cancer patients on Taxane chemo protocol will receive lidocaine i.v infusion (2 mg/kg) in 200ml saline over forty minutes with a maximum upper limit of 200 mg pre each chemotherapy session until end of the cycle. If any selected patient reported neuropathic pain (DN4 > 4) during the course of chemotherapy lidocaine (2 mg/kg) re-infused after each session. If lidocaine side effects such as circumoral numbness, twitches, metal test, tachy or bradycardia recorded at any time, lidocaine infusion will be reduced to 1mg/kg, if side effects persist, the patients will be managed accordingly as well as lidocaine infusion will be stopped and patient will be excluded from the study.
  Interventions: Drug: Lidocaine in Saline
- Group duloxetine (D) (Experimental): 20 adult breast cancer patients on chemotherapy will take oral duloxetine tablet 30 mg once per day starting from the night pre chemotherapy session until the end of cycle. If any selected patient reported neuropathic pain (DN4 > 4) during the course of chemotherapy the duloxetine dose will be adjusted to 60 mg daily till the end of the cycle. They also will receive 200 ml normal saline over forty minutes before each chemotherapy session until end of the cycle.
  Interventions: Drug: Duloxetine 30 MG

INTERVENTIONS:
Drug: Lidocaine in Saline — Lidocaine IV infusion (2 mg/kg) in 200 ml saline over forty minutes with a maximum upper limit of 200 mg pre each chemotherapy session until end of the cycle.
  Other Names: L
  Arms: Group lidocaine infusion (L)
Drug: Duloxetine 30 MG — Oral Duloxetine tablet 30 mg once per day starting from the night pre chemotherapy during the whole period of chemotherapy cycle which expected to be three month
  Other Names: D
  Arms: Group duloxetine (D)
Drug: Normal saline — 200 ml normal saline over forty minutes pre each chemotherapy session until end of the cycle.
  Other Names: C
  Arms: Group Control (C)

SUMMARY:
The aim of the study is to evaluate the effect of intravenous (IV) lidocaine versus oral duloxetine on the onset and severity of TIPN in patient with breast cancer as well as evaluation of Patients' quality of life and estimation the cell mediated immunity.

The current study is a single blinded randomized controlled study, assumed that lidocaine could prevent and reduce TIPN similar to duloxetine in patient with breast cancer.

Method of randomization: The allocation sequence was generated using permuted block randomization technique and the block size was variable. Allocation sequence/code was concealed from the person allocating the participants to the intervention arms using sealed opaque envelopes.

Primary outcome: Degree of neuropathic pain measured by neuropathy pain scale (NPS) among breast cancer patients on Taxane chemotherapy after the pretreatment with either lidocaine or duloxetine.

Secondary outcomes are: The incidence of TIPN using DN4 questionnaire and nerve conduction study and Patients' quality of life using The European Organization for Research and Treatment of Cancer (EORTC) QLQ-CIPN20 as well as the Change in serum level natural killer cell to estimate cell mediated immunity.

DETAILED DESCRIPTION:
Patients' assessment:

* Medical history (Previous diseases and medications)
* Clinical examination and laboratory investigations (according to patient' condition).
* Each patient will be informed with the study, its expected result and its possible side effects. The patients will be trained to use neuropathic pain scale (NPS). Additionally, DN4 questionnaire will be explained to all participants. IV line will be inserted for all participants. Vital signs including heart rate and mean arterial blood pressure will be measured.

The participants will be randomly allocated into three groups as follows:

* Group control (C): 20 adult breast cancer patients on Taxane chemo protocol will receive 200 ml normal saline over forty minutes pre each chemotherapy session until end of the cycle.
* Group lidocaine infusion (L): 20 adult breast cancer patients on Taxane chemo protocol will receive lidocaine IV infusion (2 mg/kg) in 200ml saline over forty minutes with a maximum upper limit of 200 mg pre each chemotherapy session until end of the cycle. If any selected patient reported neuropathic pain (DN4 > 4) during the course of chemotherapy lidocaine (2 mg/kg) re-infused after each session. If lidocaine side effects such as circumoral numbness, twitches, metal test, tachy or bradycardia recorded at any time, lidocaine infusion will be reduced to 1mg/kg, if side effects persist, the patients will be managed accordingly as well as lidocaine infusion will be stopped and patient will be excluded from the study.
* Group duloxetine (D): 20 adult breast cancer patients on chemotherapy will take oral duloxetine tablet 30 mg once per day starting from the night pre chemotherapy session until the end of cycle. If any selected patient reported neuropathic pain (DN4 > 4) during the course of chemotherapy the duloxetine dose will be adjusted to 60 mg daily till the end of the cycle. They also will receive 200 ml normal saline over forty minutes before each chemotherapy session until end of the cycle.

Measurements

Demographic features of the patients

-Age (years), Weight (kg).

Neuropathic pain characters and severity

-Intensity and characters of neuropathic pain will be measured by neuropathic pain scale (0-10cm) after each chemotherapy session which is expected to be one session every week for 12 weeks

Chemotherapy induced peripheral neuropathy

* Nerve conduction study will be performed to detect sensory peripheral neuropathy pre and immediately after the end of chemo protocol cycle.
* Detection of TIPN will be measured using DN4 questionnaire before starting chemotherapy protocol and after each chemotherapy session which is expected to be one session every week for 12 weeks

Patients' quality of life -The European Organization for Research and Treatment of Cancer (EORTC) QLQ-CIPN20 questionnaire for quality of life will be taken from patient before starting chemotherapy protocol ,one month ,two month after the treatment and at the end of treatment .

Cell mediated immunity: Natural killer cell isolation and cytotoxicity assay.

-Sample of 1ml of patients' peripheral blood will be collected on EDTA for flow cytometry to enumerate for both cytotoxic lymphocytes population (NK cells, and cytotoxic lymphocytes (ctls)). CD 56 will be used as a market for NK cells while CD8 will be used as a marker for Ctls. Cytotoxic assay will be done by measuring the release of lactate dehydrogenase (LDH) from non-viable cells (Cytotoxicity Detection kit, 630117; Clontech laboratories, Mountain View, California) according to manufacturer's instructions. Then ratio of LDH released specifically from NK cells will be carried according to the result of flow cytometry . Blood Sample will be collected at the start and the end of chemo protocol cycle of breast cancer patients.

Complications

-Any complications will occur during or after the treatment with lidocaine or duloxetine will be reported and managed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer
* at any stage,
* Taxane chemo-protocol.

Exclusion Criteria:

* Documented history of gloves and stock neuropathy.
* Alcohol abuse.
* Abnormal renal or liver function tests.
* Allergy to local anesthetics.
* Myocardial infarction within 6 months
* Profound high-grade arrhythmias.
* Patients with neurological or psychological problems.
* Diabetes Mellitus.
* History of previous chemotherapy treatment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Change in Neuropathic pain characters and severity | every week for 12 weeks (after each chemotherapy session)
  The change in intensity and characters of neuropathic pain will be measured using Neuropathy Pain Scale (NPS). It quantifies severity of neuropathic pain (0 indicates no pain, 10 indicates the most pain imaginable).

SECONDARY OUTCOMES:
Quality of life assessment using the European Organization for Research and Treatment of Cancer - Quality of life questioner - Chemotherapy induced peripheral neuropathy twenty-item scale(EORTC - QLQ - CIPN20 ). | Baseline (before starting chemotherapy protocol), one month ,two month and at 12 weeks ( end of chemotherapy cycle)
  The European Organization for Research and Treatment of Cancer (EORTC - QLQ - CIPN20) will be used to elicit patients' experience of symptoms and functional limitations related to chemotherapy induced peripheral neuropathy . It consists of 20 items with scores ranging from 1 to 4 for each item . Not at All (1), A Little (2), Quite a Bit (3), and Very much(4).
Detection of Chemotherapy induced peripheral neuropathy using sensory nerve conduction latency study . | Baseline (before starting chemotherapy protocol) then 12 weeks later ( end of chemotherapy cycle)
  Sensory nerve conduction latency study will be performed on bilateral sural and radial nerves. It test peak latency (millisecond).
Detection of Chemotherapy induced peripheral neuropathy using sensory nerve conduction amplitude study . | Baseline (before starting chemotherapy protocol) then 12 weeks later ( end of chemotherapy cycle)
  Sensory nerve conduction amplitude study will be performed on bilateral sural and radial nerves. It test amplitude (microvolt) .
Detection of Chemotherapy induced peripheral neuropathy using sensory nerve conduction velocity study . | Baseline (before starting chemotherapy protocol) then 12 weeks later ( end of chemotherapy cycle)
  Sensory nerve conduction velocity study will be performed on bilateral sural and radial nerves. It test nerve conduction velocity (meter/second).
Incidence of Taxane induced peripheral neuropathy (TIPN) using Douleur Neuropathique 4 questionnaire (DN4) | Baseline (before starting chemotherapy protocol), then every week for 12 weeks (after each chemotherapy session)
  Detection of TIPN will be measured by DN4 questionnaire .It is a clinician-administered questionnaire consisting of 10 items. Seven items related to pain quality (i.e. subjective sensory and pain descriptors) and 3 items based on the clinical examination. Scores ≥ 4/10 indicate neuropathic pain.
Change in serum level of natural killer cell to estimate cell mediated immunity | Baseline (before starting chemotherapy protocol) then 12 weeks later ( end of chemotherapy cycle)
  CD 56 will be used as a marker for NK cells while CD8 will be used as a marker for cytotoxic lymphocytes (CtLS).

CONTACTS AND LOCATIONS:
Overall Officials: Sahar A El-Karadawy, MD, Study Director — Medical Research Institute - MRI; Magda M Abo-Ollo, MD, Study Director — Medical Research Institute - MRI; Wessam Z. Alamrawy, MD, Study Director — Medical Research Institute - MRI; Yasmine N. Elwany, MD, Study Director — Medical Research Institute - MRI
Locations (1):
- Egypt Medical Research Institute, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected can be shared with other researchers in other studies as described by the main investigators. Personal data will never be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available once collected and reported in study database.
Access Criteria: All IPD collected can be shared with other researchers in other studies as described by the main investigators. Personal data will never be shared.

REFERENCES:
- [Background] Argyriou AA, Bruna J, Marmiroli P, Cavaletti G. Chemotherapy-induced peripheral neurotoxicity (CIPN): an update. Crit Rev Oncol Hematol. 2012 Apr;82(1):51-77. doi: 10.1016/j.critrevonc.2011.04.012. Epub 2011 Sep 10. PMID 21908200
- [Background] Kosharskyy B, Almonte W, Shaparin N, Pappagallo M, Smith H. Intravenous infusions in chronic pain management. Pain Physician. 2013 May-Jun;16(3):231-49. PMID 23703410
- [Background] Bril V, England JD, Franklin GM, Backonja M, Cohen JA, Del Toro DR, Feldman EL, Iverson DJ, Perkins B, Russell JW, Zochodne DW; American Academy of Neurology; American Asociation of Neuromuscular and Electrodiagnostic Medicine; American Academy of Physical Medicine and Rehabilitation. Evidence-based guideline: treatment of painful diabetic neuropathy--report of the American Association of Neuromuscular and Electrodiagnostic Medicine, the American Academy of Neurology, and the American Academy of Physical Medicine & Rehabilitation. Muscle Nerve. 2011 Jun;43(6):910-7. doi: 10.1002/mus.22092. Epub 2011 Apr 11. PMID 21484835
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] DeMarco GJ, Nunamaker EA. A Review of the Effects of Pain and Analgesia on Immune System Function and Inflammation: Relevance for Preclinical Studies. Comp Med. 2019 Dec 1;69(6):520-534. doi: 10.30802/AALAS-CM-19-000041. Epub 2019 Dec 20. PMID 31896389
- [Background] Ewertz M, Qvortrup C, Eckhoff L. Chemotherapy-induced peripheral neuropathy in patients treated with taxanes and platinum derivatives. Acta Oncol. 2015 May;54(5):587-91. doi: 10.3109/0284186X.2014.995775. Epub 2015 Mar 9. PMID 25751757
- [Background] Fallon MT. Neuropathic pain in cancer. Br J Anaesth. 2013 Jul;111(1):105-11. doi: 10.1093/bja/aet208. PMID 23794652
- [Background] Hershman DL, Lacchetti C, Dworkin RH, Lavoie Smith EM, Bleeker J, Cavaletti G, Chauhan C, Gavin P, Lavino A, Lustberg MB, Paice J, Schneider B, Smith ML, Smith T, Terstriep S, Wagner-Johnston N, Bak K, Loprinzi CL; American Society of Clinical Oncology. Prevention and management of chemotherapy-induced peripheral neuropathy in survivors of adult cancers: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jun 20;32(18):1941-67. doi: 10.1200/JCO.2013.54.0914. Epub 2014 Apr 14. PMID 24733808
- [Background] Meng J, Zhang Q, Yang C, Xiao L, Xue Z, Zhu J. Duloxetine, a Balanced Serotonin-Norepinephrine Reuptake Inhibitor, Improves Painful Chemotherapy-Induced Peripheral Neuropathy by Inhibiting Activation of p38 MAPK and NF-kappaB. Front Pharmacol. 2019 Apr 9;10:365. doi: 10.3389/fphar.2019.00365. eCollection 2019. PMID 31024320
- [Background] Mols F, Beijers T, Vreugdenhil G, van de Poll-Franse L. Chemotherapy-induced peripheral neuropathy and its association with quality of life: a systematic review. Support Care Cancer. 2014 Aug;22(8):2261-9. doi: 10.1007/s00520-014-2255-7. Epub 2014 May 1. PMID 24789421
- [Background] Pannucci CJ, Wilkins EG. Identifying and avoiding bias in research. Plast Reconstr Surg. 2010 Aug;126(2):619-625. doi: 10.1097/PRS.0b013e3181de24bc. PMID 20679844
- [Background] Rivera DR, Ganz PA, Weyrich MS, Bandos H, Melnikow J. Chemotherapy-Associated Peripheral Neuropathy in Patients With Early-Stage Breast Cancer: A Systematic Review. J Natl Cancer Inst. 2018 Feb 1;110(2):djx140. doi: 10.1093/jnci/djx140. PMID 28954296
- [Background] Saarto T, Wiffen PJ. Antidepressants for neuropathic pain. Cochrane Database Syst Rev. 2007 Oct 17;2007(4):CD005454. doi: 10.1002/14651858.CD005454.pub2. PMID 17943857
- [Background] Shimozuma K, Ohashi Y, Takeuchi A, Aranishi T, Morita S, Kuroi K, Ohsumi S, Makino H, Katsumata N, Kuranami M, Suemasu K, Watanabe T, Hausheer FH. Taxane-induced peripheral neuropathy and health-related quality of life in postoperative breast cancer patients undergoing adjuvant chemotherapy: N-SAS BC 02, a randomized clinical trial. Support Care Cancer. 2012 Dec;20(12):3355-64. doi: 10.1007/s00520-012-1492-x. Epub 2012 May 15. PMID 22584733
- [Background] Skljarevski V, Desaiah D, Liu-Seifert H, Zhang Q, Chappell AS, Detke MJ, Iyengar S, Atkinson JH, Backonja M. Efficacy and safety of duloxetine in patients with chronic low back pain. Spine (Phila Pa 1976). 2010 Jun 1;35(13):E578-85. doi: 10.1097/BRS.0b013e3181d3cef6. PMID 20461028
- [Background] Starobova H, Vetter I. Pathophysiology of Chemotherapy-Induced Peripheral Neuropathy. Front Mol Neurosci. 2017 May 31;10:174. doi: 10.3389/fnmol.2017.00174. eCollection 2017. PMID 28620280
- [Background] Wang YJ, Chan YN, Jheng YW, Wu CJ, Lin MW, Tseng LM, Tsai YF, Liu LC. Chemotherapy-induced peripheral neuropathy in newly diagnosed breast cancer survivors treated with taxane: a prospective longitudinal study. Support Care Cancer. 2021 Jun;29(6):2959-2971. doi: 10.1007/s00520-020-05796-0. Epub 2020 Oct 6. PMID 33025227
- [Background] Westbom C, Thompson JK, Leggett A, MacPherson M, Beuschel S, Pass H, Vacek P, Shukla A. Inflammasome Modulation by Chemotherapeutics in Malignant Mesothelioma. PLoS One. 2015 Dec 21;10(12):e0145404. doi: 10.1371/journal.pone.0145404. eCollection 2015. PMID 26689911
- [Background] Willison HJ, Winer JB. Clinical evaluation and investigation of neuropathy. J Neurol Neurosurg Psychiatry. 2003 Jun;74 Suppl 2(Suppl 2):ii3-ii8. doi: 10.1136/jnnp.74.suppl_2.ii3. No abstract available. PMID 12754322
- [Background] Zhi WI, Chen P, Kwon A, Chen C, Harte SE, Piulson L, Li S, Patil S, Mao JJ, Bao T. Chemotherapy-induced peripheral neuropathy (CIPN) in breast cancer survivors: a comparison of patient-reported outcomes and quantitative sensory testing. Breast Cancer Res Treat. 2019 Dec;178(3):587-595. doi: 10.1007/s10549-019-05416-4. Epub 2019 Aug 27. PMID 31456070
- [Background] Chatila N, Pereira B, Maarrawi J, Dallel R. Validation of a New Arabic Version of the Neuropathic Pain Diagnostic Questionnaire (DN4). Pain Pract. 2017 Jan;17(1):78-87. doi: 10.1111/papr.12419. Epub 2016 Feb 20. PMID 26895970
- [Background] Galer BS, Jensen MP. Development and preliminary validation of a pain measure specific to neuropathic pain: the Neuropathic Pain Scale. Neurology. 1997 Feb;48(2):332-8. doi: 10.1212/wnl.48.2.332. PMID 9040716
- [Background] Schulz KF, Grimes DA. Allocation concealment in randomised trials: defending against deciphering. Lancet. 2002 Feb 16;359(9306):614-8. doi: 10.1016/S0140-6736(02)07750-4. PMID 11867132
- [Background] Schulz KF, Grimes DA. Generation of allocation sequences in randomised trials: chance, not choice. Lancet. 2002 Feb 9;359(9305):515-9. doi: 10.1016/S0140-6736(02)07683-3. PMID 11853818
- [Background] van Haren F, van den Heuvel S, Radema S, van Erp N, van den Bersselaar L, Vissers K, Steegers M. Intravenous lidocaine affects oxaliplatin pharmacokinetics in simultaneous infusion. J Oncol Pharm Pract. 2020 Dec;26(8):1850-1856. doi: 10.1177/1078155220905011. Epub 2020 Feb 19. PMID 32075507
- [Background] Perez C, Galvez R, Huelbes S, Insausti J, Bouhassira D, Diaz S, Rejas J. Validity and reliability of the Spanish version of the DN4 (Douleur Neuropathique 4 questions) questionnaire for differential diagnosis of pain syndromes associated to a neuropathic or somatic component. Health Qual Life Outcomes. 2007 Dec 4;5:66. doi: 10.1186/1477-7525-5-66. PMID 18053212
- [Result] Areti A, Yerra VG, Naidu V, Kumar A. Oxidative stress and nerve damage: role in chemotherapy induced peripheral neuropathy. Redox Biol. 2014 Jan 18;2:289-95. doi: 10.1016/j.redox.2014.01.006. eCollection 2014. PMID 24494204
- [Derived] Abouelmagd GMT, El-Karadawy SA, Abo-Ollo MM, Elwany YN, Mohamed ER, El-Amrawy WZ. Lidocaine Infusion Versus Duloxetine for Prevention and Management of Taxane-Induced Peripheral Neuropathy among Breast Cancer Patients-A Randomized Controlled Study. Pain Physician. 2023 Sep;26(5):E497-E507. PMID 37774185